CLINICAL TRIAL: NCT03428386
Title: Single-Anastomosis Plication Ileal Bypass in Treatment of Morbid Obesity: a Pilot Study
Brief Title: Single-Anastomosis Plication Ileal Bypass for Morbid Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mansourau46
Record Dates: First submitted 2018-02-04; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastric plication ileal bypass (Experimental): single-anastomosis plication ileal bypass
  Interventions: Procedure: Gastric plication ileal bypass

INTERVENTIONS:
Procedure: Gastric plication ileal bypass — laparoscopic plication of the greater curvature of the stomach then the duodeno-jejunal junction is identified and 300 cm is measured downwards. The selected loop will be ascended without division of the greater omentum, and a stapled isoperistaltic side-to-side to the anterior wall of the antrum of the stomach just 3 cm away from the pylorus with a linear stapler charged with a green cartridge, the diameter of ileal antrum anastomosis is not exceeding 3 cm in diameter. The staple defect is closed with a two-layer running 3/0 polyglactin suture

SUMMARY:
The present study aims to explore the impact of combining laparoscopic greater curvature plication with a single gastro-ileal anastomosis in the same manner of single anastomosis sleeve ileal bypass on weight loss and postoperative complications. The objective of this combined procedure is to reduce the high intraluminal pressure that results after laparoscopic greater curvature plication owing to reduced intraluminal space which can lead to suture line leakage, vomiting, and gastroesophageal reflux disease. Another objective is to add a malabsorptive element to the restrictive effect of laparoscopic greater curvature plication and to induce early satiety in patients by distention of the distal bowel with nutrients immediately after meals, similar to the way that single anastomosis sleeve ileal bypass works.

DETAILED DESCRIPTION:
The present study aims to explore the impact of combining laparoscopic greater curvature plication with a single gastro-ileal anastomosis in the same manner of single anastomosis sleeve ileal bypass on weight loss and postoperative complications. The objective of this combined procedure is to reduce the high intraluminal pressure that results after laparoscopic greater curvature plication owing to reduced intraluminal space which can lead to suture line leakage, vomiting, and gastroesophageal reflux disease. Another objective is to add a malabsorptive element to the restrictive effect of laparoscopic greater curvature plication and to induce early satiety in patients by distention of the distal bowel with nutrients immediately after meals, similar to the way that single anastomosis sleeve ileal bypass works.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders aging between 18 and 60 years with morbid obesity will be included to the study

Exclusion Criteria:

* Patients with secondary obesity due to endocrine disorders
* patient unfit for general anesthesia.
* patients who had not attempted non-surgical weight loss treatment in the past
* patients with psychological conditions that influence his/her perception of the study protocol
* patients with previous surgery for morbid obesity

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
weight loss | 6 months
  Percentage of excess weight loss at 6 months after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D., Principal Investigator — Mansoura University Hospital
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No